CLINICAL TRIAL: NCT04479644
Title: A Phase 1 Randomized, Single-blind, Placebo-controlled, Single Ascending Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Human Monoclonal Antibody, BRII-198 Administered Intravenously to Healthy Adult Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics Study of Human Monoclonal Antibody BRII-198
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Collaborators: TSB Therapeutics (Beijing) CO.LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRII-198-001
Record Dates: First submitted 2020-07-14; First posted 2020-07-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19 phase I; monoclonal antibody
MeSH Terms: conditions — COVID-19 | interventions — romlusevimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): BRII-198 dose level 1 or placebo
  Interventions: Drug: BRII-198; Drug: Placebo
- Cohort 2 (Experimental): BRII-198 dose level 2 or placebo
  Interventions: Drug: BRII-198; Drug: Placebo
- Cohort 3 (Experimental): BRII-198 dose level 3 or placebo
  Interventions: Drug: BRII-198; Drug: Placebo

INTERVENTIONS:
Drug: BRII-198 — BRII-198 given intravenously
Drug: Placebo — Placebo given intravenously

SUMMARY:
This is a phase 1 study in which healthy adult volunteers will receive BRII-198 or placebo and will be assessed for safety, tolerability, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 49 years of age inclusive;
* Body weight ≤100 kg and body mass index (BMI) within the range of 19.0-24.0kg/m2 (inclusive);
* Male or female;

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation;
* A history of significant hypersensitivity, intolerance, or allergy to any drug compound;
* History of alcohol or other substance abuse;

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) by CTCAE v5.0 | up to 24 weeks
Proportion of subjects with SAEs | up to 24 weeks
Proportion of subjects with infusion-related reactions | up to 24 weeks
Proportion of subjects with hypersensitivity reactions | up to 24 weeks

SECONDARY OUTCOMES:
Serum Concentration of BRII-198 | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhang, Study Director — TSB Therapeutics (Beijing) CO.LTD
Locations (1):
- Investigative Site, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hao X, Zhang Z, Ma J, Cheng L, Ji Y, Liu Y, Zhao D, Zhang W, Li C, Yan L, Margolis D, Zhu Q, Zhang Y, Zhang F. Randomized, placebo-controlled, single-blind phase 1 studies of the safety, tolerability, and pharmacokinetics of BRII-196 and BRII-198, SARS-CoV-2 spike-targeting monoclonal antibodies with an extended half-life in healthy adults. Front Pharmacol. 2022 Sep 6;13:983505. doi: 10.3389/fphar.2022.983505. eCollection 2022. PMID 36147329
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343